CLINICAL TRIAL: NCT05970107
Title: A Prospective Randomized Trial of Axillary Node Dissection With or Without Lymphaticovenous Bypass (LVB) in Node Positive Breast Cancer Patients
Brief Title: Axillary Node Dissection w or w/o LVB in Node Positive Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2123
Record Dates: First submitted 2023-06-13; First posted 2023-08-01 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Node-positive Breast Cancer
Keywords: Prophylactic Lymphaticovenous Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALND + LVB (Experimental): The prophylactic LVB cohort will undergo ALND plus ARM and immediate lymphatic reconstruction with lymphaticovenous bypass (LVB). During the ALND, axillary reverse mapping will be used to visualize the lymphatics draining into the axilla, to aid in preserving the draining lymphatic vessels for anastomosis in LVB.
  Radiation therapy will be administered as determined by the treating radiation oncologist.
  Interventions: Procedure: Axillary Lymph Node Dissection; Procedure: Axillary Reverse Mapping; Procedure: Lymphaticovenous Bypass
- ALND without LVB (Active Comparator): Patients in the ALND alone cohort will undergo ALND plus ARM
  Radiation therapy will be administered as determined by the treating radiation oncologist.
  Interventions: Procedure: Axillary Lymph Node Dissection; Procedure: Axillary Reverse Mapping

INTERVENTIONS:
Procedure: Axillary Lymph Node Dissection — ALND happens after cancer cells are found during a sentinel lymph node biopsy.
  ALND can remove lymph nodes located above, below or directly underneath a muscle that runs along the side of the upper chest.
  Other Names: ALND
Procedure: Axillary Reverse Mapping — Axillary reverse mapping (ARM) is a technique where blue dye is injected into the upper arm at surgery, allowing direct visualization of arm lymphatics and nodes during ALND
  Other Names: ARM
Procedure: Lymphaticovenous Bypass — Lymphaticovenous bypass/anastomosis (LVB/LVA) involves supramicrosurgery in which the blocked lymphatic vessel of an affected limb is connected to a nearby vein with the aid of ultra-fine instruments and a powerful operating microscope.
  Other Names: LVB
  Arms: ALND + LVB

SUMMARY:
Lymphedema is a devastating complication of breast cancer surgery that decreases the quality of life of up to 40% of breast cancer survivors. Most lymphedema in breast cancer patients is because lymphatics shared between the axilla and the arm are sacrificed during axillary lymph node dissection (ALND) surgery, which removes an average of 15 lymph nodes in node positive patients. CCF's breast cancer plastic microvascular surgeons and breast surgical oncologists have collaborated to refine a surgical technique known as LVB that may be used either as a preventive measure (prophylactic LVB) or as a therapeutic intervention (therapeutic LVB). Lymphatic reconstruction with LVB may be an improvement to the current standard of care for node positive breast cancer patients undergoing ALND.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed axillary node positive unilateral breast cancer and may be female or male.
* Subjects must have received no prior surgical interventions to the axilla except for core needle biopsy or sentinel node biopsy within 30 days of the planned axillary node dissection.
* Age >18 years. Children are excluded from this study since breast cancer is quite rare in children.
* ECOG Performance status 0 or 1
* Subjects must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine within normal institutional limits
* Subjects must have at least one suitable lymphatic and one suitable vein amenable to lymphovenous bypass anastomosis.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Patients may be treated with adjuvant or neoadjuvant therapies at the discretion of the treating medical oncologist
* Patients may be treated with adjuvant radiation therapy at the discretion of the treating radiation oncologist.
* Patients may be treated with either mastectomy or breast conserving surgery at the discretion of the treating surgical oncologist.
* In order to complete the Lymph-ICF-UL questionnaire, participants must be able to speak and/or read English.
* Healthy controls include women aged 18-75 without a current or past history of breast cancer or lymphedema who are willing to undergo blood draw.

Exclusion Criteria:

* Contraindication to ICG as a) iodine hypersensitivity, b) renal failure, c) uremia and d) on dialysis.
* Subjects receiving any prior surgical treatment or radiation to the axilla prior to protocol enrollment (except sentinel node biopsy within the past 30 days).
* Subjects with known regional cervical or supraclavicular nodal disease or distant metastatic disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to isosulfan blue dye or other agents used in this study.
* History of pre-existing lymphedema or measured lymphedema at baseline upon study enrollment
* BMI greater than or equal to 40.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of pulmonary embolism or deep venous thrombosis
* Patients must not be on anticoagulant therapy with warfarin, clopidogrel (Plavix), apixavan (Eliquis), heparin, low molecular weight heparin, rivaroxaban (Xarelto), ticlodipine (Ticlid), fonduparinux (Arixtra) with the exception of routine heparin flushes to a portacath.
* Patients treated with sentinel lymph node biopsy only without ALND
* Arteriovenous fistula or the presence of an indwelling peripherally inserted central catheter (PICC line), or the presence of a central venous line or portacath in the ipsilateral arm.
* ECOG performance status of 2 or higher.
* Pregnant or breast-feeding women are excluded from the study given that it is unknown whether isosulfan blue can cause fetal harm and it is desirable to limit anesthesia time in this population
* Less than 18 years of age or greater than 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 4 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 8 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 12 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 16 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 20 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 24 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Objective Criteria | At month 27 post treatment
  This is defined as a diagnosis of lymphedema by at least three of the four objective measurements performed serially every four months after baseline.
  The four diagnostic measurements to be performed at baseline and then every four months during the study timeframe are: a) Limb measurements; b) 3D Infrared optoelectronic volumetry (Perometer); c) Bioimpedence Spectroscopy (LDEX); d) LymphaTech handheld 3D scan.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 4 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 8 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 12 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 16 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 20 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 24 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.
Rate of lymphedema onset after prophylactic LVB-Subjective Criteria | At month 27 post treatment
  The patient-reported outcomes survey Lymph-ICF-UL will be used to compare subjective symptoms of lymphedema to the four diagnostic measurements to determine which is the most sensitive and evaluate the concordance of these tests.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Lang, MD, FACS, Principal Investigator — Cleveland Clinic Foundation: Digestive Disease & Surgery Institute